CLINICAL TRIAL: NCT01159184
Title: Stressors, Coping Methods and Social Support in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ju-Ying Jiang, Attending physician, Far Eastern Memorial Hospital
Other Study IDs: 098083-3
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes
Keywords: stress; coping methods; social support; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The increasing prevalence of diabetes brought great burden to health status of the investigators population. It is meaningful to investigate the stressor, stress perceived, social support and coping methods in diabetic population in order to provide appropriate assistance to these patients. This study will recruit diabetes patients from out-patient-department and they are invited to complete a questionnaire. The contents of the questionnaire including stress experienced, stress perceived, social support and coping methods. The investigators purpose is to find out the impact of these factors on glycemic controlled and their life quality. The results will be useful to diabetes care team when health education is delivered to patient.

DETAILED DESCRIPTION:
Type 2 diabetes patient aged 30-80 y/o under oral hypoglycemic agents with clear conscious enable to answer questions properly who regularly follow up at our metabolism clinic is eligible. Patients are asked to complete a questions containing basic personal information, diabetes coping method Chinese version (DCM-C)questionnaire, social support and perceived stress scale.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Aged 30-80 year old
3. under oral hypoglycemic agents
4. clear consciousness

Exclusion Criteria:

1. Type 1 diabetes
2. Age below 30 and above 80
3. Insulin use
4. Conscious not clear

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Type 2 diabetes
  2. Aged 30-80 year old
  3. under oral hypoglycemic agents
  4. clear consciousness
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ju Ying Jiang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan